CLINICAL TRIAL: NCT06239844
Title: Navigating Together for Equitable Asthma Management for Children in Families Who Communicate in Languages Other Than English (Nav-TEAM)
Brief Title: Navigating Together for Equitable Asthma Management for Children in Families Who Communicate in Language Other Than English
Acronym: Nav-TEAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 23-1544
Record Dates: First submitted 2023-11-06; First posted 2024-02-02 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Asthma in Children

STUDY DESIGN:
Intervention Model Description: The proposed study builds on a successful local model of asthma navigation and care coordination to support meeting social determinants of health (SDOH) needs using a lay health worker model that has improved asthma outcomes among urban racial/ethnic minority school children. This model is currently being disseminated via community-engaged processes to select school districts across Colorado. Community advisory board members from that initiative identified increasing language inclusivity as a priority in program dissemination.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nav-Team (Experimental): Participants in this arm will receive additional assistance related to asthma, and will participate in encounters over the subsequent 9 months
  Interventions: Other: Experimental: Nav-Team
- Non-Nav-Team (No Intervention): Participants in this arm will participate in surveys but will receive no navigation assistance.

INTERVENTIONS:
Other: Experimental: Nav-Team — Participants in this arm will receive additional assistance related to asthma, log encounters, complete surveys.
  Arms: Nav-Team

SUMMARY:
The Nav-Team study reviews how well the asthma navigators/coordinator program can improve the lives of asthmatic children, and their caregivers, by providing additional assistance and education. Aim 1 of the study will partner with immigrant serving community organizations to hold meetings that will help tailor the programs. Aim 2 of the study looks at data to help see if the program is working to help children and their caregivers. Aim 2a looks at difference in emergency department use between families that did not use the Nav-Team program and those that did. Aim 2b reviews how well the Nav-Team program did with reaching and connecting with the asthma child and caregiver community. Aim 2b, also reviews the costs of the program, how well the program did will sticking to the program goals, and how well the staff was able to keep up with providing education and help.

DETAILED DESCRIPTION:
Children in families with healthcare communication in a language other than English are at increased risk of poor asthma care and worse asthma outcomes compared to those without a language barrier. As the most common chronic childhood disease, asthma causes substantial family- and patient-level burden as well as economic impact. Caregivers of children with asthma whose healthcare communication is in languages other than English (LOE) are more likely to report poor asthma care experiences, less use of recommended asthma management practices, and higher hospitalization rates compared to children with caregivers with English healthcare communication. A focus on improving asthma care specifically for families who communicate in LOE is needed to address such disparities.

Asthma navigators play a key role in asthma education and care coordination, resulting in improved asthma outcomes, particularly for low-income and racial/ethnic minority children but studies have not focused on children in LOE families. The proposed study builds on a successful local model of asthma navigation and care coordination to support meeting social determinants of health (SDOH) needs using a lay health worker model that has improved asthma outcomes among urban racial/ethnic minority school children. This model is currently being disseminated via community-engaged processes to select school districts across Colorado. Community advisory board members from that initiative identified increasing language inclusivity as a priority in program dissemination. However, school feasibility concerns and limited opportunities for cultural and language tailoring prevent focusing on this priority. Addressing these barriers, the Navigating Toward Equitable Asthma Management Program (Nav-TEAM) is an adaptation of evidence-based asthma navigation specifically for children in families who communicate in LOE.

Nav-TEAM will include core components of evidence-based asthma navigation/care coordination through a different implementation approach and via specific tailoring for LOE families. Children with asthma and their families will be connected to Nav-TEAM via their healthcare provider rather than the school. Nav-TEAM encounters will take place via telehealth because frequent asthma care in clinic can be difficult for families, and home visits present coordination challenges and increased costs. While emerging research points to inequitable reach of telehealth for LOE patients/families, the telehealth program at the proposed study health system, is committed to equity via integrated interpretation and continuous improvement to increase use with LOE families informed by research partnerships to assess telehealth equity.

Use of lay health workers to provide asthma education and care coordination is a well-established effective intervention. Nav-TEAM will build on the successes of school and home-visiting programs affiliated with the study health system, Children's Hospital Colorado (CHCO) with a novel focus on reaching LOE families. As with existing CHCO asthma navigation programs, Nav-TEAM will align with EXHALE, the Centers for Disease Control and Prevention National Asthma Control Program compilation of asthma management strategies that have been proven to reduce asthma-related ED visits, hospitalization, and healthcare costs. EXHALE strategies include EDUCATION on asthma -self-management, X-TINGUISHING smoking and exposure to secondhand smoke, Home Visits, ACHIEVEMENT of guidelines-based medical management, LINKAGES and coordination of care across settings, ENVIRONMENTAL policies & best practices to reduce asthma triggers.

When will Nav-TEAM Encounters occur and what will take place during encounters? Families will participate in the Nav-TEAM intervention for 9 months which is similar to the length of school- and home-based programs. There will be scheduled Nav-TEAM encounters with additional encounters to follow-up any asthma-related clinic, ED or hospital visits. We expect most patients will complete ≈6 encounters based on current utilization patterns. Encounters will follow an intervention guide used in existing programs with some adapted elements based on Aim 1 feedback and tailoring. There will be the availability to schedule Nav-TEAM encounters during evening hours and to accommodate families' work schedules.

The overall scientific goals of this community-engaged study are to: evaluate the effectiveness of Nav-TEAM on pediatric asthma outcomes for 320 children whose families communicate in LOE, evaluate implementation outcomes, and assess cost and contextual factors to support sustained implementation, scale up and scale out. The study will be implemented in a large primary care clinic serving primarily Medicaid-insured children and in subspecialty pediatric pulmonary clinics using the Practical Robust Implementation and Sustainability Model (PRISM) - inclusive of RE-AIM (Reach, Effectiveness, Adoption, Implementation Maintenance outcomes with an equity lens- as the guiding Dissemination & Implementation Science framework.

ELIGIBILITY:
eria for Nav-TEAM Intervention Dyads include:

* Child aged 4-12 years.
* Child with persistent asthma (defined by currently prescribed controller medication).
* Parent/legal guardian who is at least 18 years old.

Exclusion criteria for Nav-TEAM Intervention Dyads include:

* Child aged under 4 and over 12 years of age.
* Child with no persistent asthma (defined by currently prescribed controller medication).
* Parent/legal guardian who is under 18 years old.
* Any parent/legal guardian whose preferred spoken language is English.
* Child requires additional continuous respiratory support (e.g,. tracheostomy with home ventilation, continuous daytime oxygen).
* Child is enrolled in another study health system associated asthma navigation program (e.g. school or home-visiting programs).
* Spoken non-English preferred healthcare language of parent/legal guardian.
* Child does NOT require additional continuous respiratory support (e.g., nighttime use of Continuous positive airway pressure machine for obstructive sleep apnea would be eligible).
* Child does NOT have a complex medical/genetic condition that affects swallowing or lung function (e.g. g-tube with aspiration, cystic fibrosis)
* Child is NOT enrolled in another study health system associated asthma navigation program (e.g. school or home-visiting programs).

Ages: 4 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2025-03-21 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Asthma-related emergency department (ED) utlization | 12 months
  Count of asthma-related ED visits based on EHR ED encounters and corresponding encounter diagnosis codes during the trial period

SECONDARY OUTCOMES:
Parent-reported asthma-related ED utilization | 12 months
  Sum of counts of asthma-related ED use based on parent-report. Asthma-related ED use in the past 3 months will be assessed via parent survey. At 3, 6,9, and 12 months this will be determined via a question on the Asthma Care Questionnaire (ACQ. The ACQ will be delivered via text-link for most participants. At 15 months parents will report asthma-related ED use in the past 3 months on the follow-up survey.
Asthma hospitalization | 12 months
  Count of asthma-related hospitalizations based on EHR ED encounters and corresponding encounter diagnosis codes
Parent-reported asthma-related hospitalization | 12 months
  Sum of counts of asthma-related hospitalization based on parent-report. Asthma-related hospitalization in the past 3 months will be assessed via parent survey. This will be determined at 3, 6, 9, and 12 months via an ACQ question. The ACQ will be delivered via text-link for most participants. At 15 months parents will report asthma-related hospitalization the past 3 months on the follow-up survey.
Asthma Exacerbations | 12 months
  % of patients with an oral steroid burst during the trial period. We define the need for oral steroids as an asthma exacerbation. Steroid bursts in the past 3 months will be assessed via parent survey. This will be determined at 3, 6, 9, and 12 months via an ACQ question. The ACQ will be delivered via text-link for most participants. At 15 months parents will report steroids bursts in the past 3 months on the follow-up survey.
Asthma Control | 12 months
  % of Asthma Control Test scores in the complete/well-controlled range (Score >19) Sum of counts of child missed school days based on parent-report. The Asthma Control Test will be administered at 3, 6, 9, and 12 months as part of the ACQ. The ACQ will be delivered via text-link for most participants. At 15 months parents will complete an additional Asthma Control Test on the follow-up survey.
Missed School Days | 12 months
  Sum of counts of child missed school days based on parent-report. Missed school days in the past 3 months will be assessed via parent survey. This will be determined at 3, 6, 9, and 12 months via an ACQ question. The ACQ will be delivered via text-link for most participants. At 15 months parents will report missed school days the past 3 months on the follow-up survey.
Missed Work Days | 12 months
  Sum of counts of parent missed work days based on parent-report. Missed work days in the past 3 months will be assessed via parent survey. This will be determined at 3, 6, 9, and 12 months via an ACQ question. The ACQ will be delivered via text-link for most participants. At 15 months parents will report missed work days the past 3 months on the follow-up survey.
General child health | 12 months
  Assessed via the PROMIS® Pediatric Global Health questionnaire which will be included in the follow-up survey
Child asthma-related quality of life | 12 months
  Assessed via the the PROMIS® Asthma Impact Scale which will be included in the follow-up survey.
Parent asthma-related quality of life | 12 months
  Assessed via the Pediatric Asthma Caregiver's Quality of Life Questionnaire which will be included in the follow-up survey.
Parent asthma self-efficacy | 12 months
  Assessed via the Parental Asthma Management Self-Efficacy Scale which will be included in the follow-up survey

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States